CLINICAL TRIAL: NCT05957224
Title: An Intervention Comparing Changes in the Plasma Glucose Profile Over a Three-hour Timespan in Persons With T2DM Following Caribbean Shake vs Glucerna Intake: A Double Blinded, Cross-over Design
Brief Title: Differences in Postprandial Glucose Changes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of The West Indies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: SHIFT
Record Dates: First submitted 2023-07-05; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus, Type II; Overweight or Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: There is a one-week washout period between intake of the two shakes.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants will be blinded to the intervention as the shakes will be given in unmarked containers - however as the flavours are very different it is likely that participants will be able to tell them apart. Data analysts will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shake 1 then Shake 2 (Experimental): Participants will consume 1 bottle of shake 1 and take their normal morning medications. After this 3ml blood samples will be taken via the cannula at 30mins, 60mins and 120 mins post meal. During the waiting period between phlebotomy, a sensory analysis questionnaire which asks participants to rate the taste, appearance, texture and smell of the product. After a 1-week washout period, the entire protocol will be repeated using Shake 2.
  Interventions: Other: Shake 1 then Shake 2
- Shake 2 then Shake 1 (Experimental): Participants will consume 1 bottle of Shake 2 and take their normal morning medications. After this 3ml blood samples will be taken via the cannula at 30mins, 60mins and 120 mins post meal. During the waiting period between phlebotomy, a sensory analysis questionnaire which asks participants to rate the taste, appearance, texture and smell of the product. After a 1-week washout period, the entire protocol will be repeated using Shake 1.
  Interventions: Other: Shake 2 then Shake 1

INTERVENTIONS:
Other: Shake 1 then Shake 2 — Oral administration of Caribbean low-calorie meal-replacement shake then commercial low-calorie meal-replacement shake
  Arms: Shake 1 then Shake 2
Other: Shake 2 then Shake 1 — Oral administration of commercial low-calorie meal-replacement shake then Caribbean low-calorie meal-replacement shake
  Arms: Shake 2 then Shake 1

SUMMARY:
Following a meal, in nondiabetic individuals, blood glucose rises to peak at 1hr and returns to baseline in 2 - 3 hours. In T2DM, this peak is higher and prolonged. Meal plans for persons with T2DM should comprise evenly spaced, complex carbohydrate portions in order to avoid post-prandial glucose spikes. Researchers have developed an expanded line of Caribbean-flavoured, low-calorie meal-replacement shakes which have been formulated to match the macronutrient and caloric content of a commercially available brand. In this trial investigators aim to (1) examine the change in glucose levels post intake of Caribbean vs the commercially available brand and (2) to conduct a comparative sensory analysis of the two shakes.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of T2DM for any length of time,
2. last HbA1C (within the last 6 months) of < / = 8%

Exclusion Criteria:

1. On insulin for any length of time

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Change in plasma glucose concentration post oral intake of shake | 30 minutes, 60 minutes and 120 minutes post oral intake of shake

SECONDARY OUTCOMES:
Sensory analysis of taste, texture, smell and appearance of shakes | within 1hour post oral intake of shake
  measured on a 5-point hedonic scale